CLINICAL TRIAL: NCT04741932
Title: Interprofessional Dementia Care: Redistribution of Tasks Between Physicians and Qualified Nurses in Primary Care
Brief Title: Interprofessional Dementia Care
Acronym: InDePendent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Medicine Greifswald (Other); University Medicine Rostock (Unknown); GNEF Gesundheitsnetz Frankfurt am Main eG (Unknown); Haffnet Management GmbH (Unknown); Demenznetzwerk Uckermark e.V. (Unknown); Techniker Krankenkasse (Other); AOK Nordost (Industry); Federal Joint Committee (Other Government)
Responsible Party: Principal Investigator, Wolfgang Hoffmann, Group Leader and Site Speaker, German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01NVF18034
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Dementia; Nurse's Role; Nurse Physician Relations
Keywords: Dementia; Dementia Care; Caregiver of people with dementia; Unmet needs; Medical management
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Special qualified nurses with an extended nursing role (Dementia Care Manager) record all nursing, medical, drug, psychosocial and social care needs using an IT-based care management system and then implement them over a period of six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention)
- Intervention (Experimental)
  Interventions: Other: Dementia Care Management (DCM)

INTERVENTIONS:
Other: Dementia Care Management (DCM) — A computerized "Information and Care Management System" (IMS) will identify unmet nursing, medical, psychosocial and social needs of the PwD and its informal caregiver. Based on this data, the IMS generates suggestions for interventions: The DCM in cooperation with the general practitioner (GP) develops an individual treatment and care plan that is tailored to the needs of the PwD and its caregiver. The DCM will initiate the implementation of respective actions and monitor the status of implementation. Therefore, the DCMs are supposed to take on activities that were previously usually performed by doctors (redistribution of tasks between physicians and qualified nurses in primary care).
  Arms: Intervention

SUMMARY:
Currently, around 1.7 million people with dementia live in Germany. The number of new cases per year is estimated to be around 244,000. At this time, no curative treatment for dementia exists. The progression of the disease results in high needs for care. Only a minority among People with Dementia (PwD) receive needs-based treatment and directive-compliant care. Previous studies found that more than 95% of PwD have an open need for care. The increase in chronically and multimorbid impaired patients leads to an increased number of patients in primary care. Particularly in rural regions, innovative care concepts based on a redistribution of tasks between specialized nurses and doctors could help to guarantee high-value care at all times. Nursing care can be expanded with regards to tasks and competencies, which is thought to increase the attractiveness of the nursing profession. Unfortunately, there are currently no scientific studies on the effectiveness and impact of such care concepts in Germany.

The Aim of this study is to implement a structured care concept for the reallocation of tasks between general practitioners (GPs) and nurses and to evaluate its effectiveness on the living and care situation of people with dementia living at home. "InDePendent" is a multicenter, cluster-randomized, controlled intervention study with a waiting-control group. Randomization is carried out at the level of the participating GPs in a ratio of 1:2 (intervention group : waiting-control group).

DETAILED DESCRIPTION:
Previous studies found that PwD treated by primary care physicians on average have 8.8 (± 5.04; range = 0-31) unmet care needs, mainly related to nursing care (38%) and drug therapy (15%). PwD had additional needs for daily activities, social participation and showed a high level of psychological stress. The number of unmet care needs is more dependent on the physical limitations than on the cognitive impairments. The progression of dementia is therefore associated with an increase in open and unmet care needs and a reduced opportunity to recognize these needs in the primary care setting and to address them appropriately. At this time, no curative treatment for dementia exists. Thus, innovative models of high-value care have to be found in order to enable PwD to live an independent, self-determined life with a high quality of life for as long as possible. The increasing burden of disease associated with an increase in prevalence of dementia is associated with high health expenditures, which puts additional pressure on health care systems. From a health economical perspective the minimization of supply deficits and open needs of care are crucial aspects to avoid or delay a cost-intensive transfer to an inpatient facility. The overall goal of the InDePendent project is to improve the living and care situation of PwD and their relatives at home. Following this aim, an innovative redistribution of tasks between general practitioners and specialized nurses for dementia patients will be implemented and evaluated. In addition, the specialized nurses will be trained for cross-sector as well as cross-professional dementia care management (DCM), by acquisition of specific competencies to carry out medical tasks in delegation and substitution. Collaborating Dementia Networks and GP clinics will serve as the units of randomization and determine the patients' group status (control or intervention group). The GPs will systematically screen the patients for eligibility to participate in the study during routine care (eligibility criteria for screening: age ≥70 years, living at home). Patients will be screened using the validated DemTect questionnaire (eligibility for study participation: <9 points). In case of a positive screening or an existing dementia diagnosis, potential participants will receive detailed information about the study including a study-information sheet from their GP, be invited to participate and asked to provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 70+ years
* PwD lives at home
* existing dementia diagnosis or screening result of DemTect <9
* caregiver: main caregiver of a PwD (Hauptversorgungsperson)

Exclusion Criteria:

- not able to provide written consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 471 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of unmet needs (CANE) | 6 months after baseline assessment
  The CANE questionnaire (Camberwell Assessment of Need for the Elderly, Stein et al., 2019) will be used to assess participants' and their relatives' unmet needs in group comparison between IG compared to the CG. The CANE comprises 27 areas of daily life for assessing the physical, psychological, social and environmental needs of older people.
  There are two versions of the CANE for both participant and caregiver.

SECONDARY OUTCOMES:
Quality of life (Qol-AD) | 6 months after baseline assessment
  The Quality of life in Alzheimer's Disease (Qol-AD; Logsdon et al. 2002) will be used to assess participants' quality of life. The instrument contains 13 items. Each item is rated on a four point likert scale, in which 1 stands for being poor and 4 being excellent. Result is a sum of all 13 items from 13 to 52. Higher numbers indicate higher quality of life.
Health status (EQ-5D-5L) | 6 months after baseline assessment
  The EQ-5D-5L instrument (Janssen et al. 2013) will be used to assess participants' health status, quality of life and for the health economic evaluation. The instrument contains 5 dimensions and one score from 0 to 100 to assess participants' current health status. Each of the 5 dimensions (Mobility, Self-care, Usual activities, Pain/Discomfort, Anxiety/ Depression) are rated on a five point likert scale. Result of the EQ-5D-5L is an individual health index.
Costs of informal care (Resource Utilization in Dementia) | 6 months after baseline assessment
  Informal care is an essential part of society's resource consumption and the costs of dementia care. For the health economic evaluation the RUD (Resource Utilization in Dementia Questionnaire, Wimo, Jonsson & Zbrozek, 2010) will be used to determine the supply costs and the informal care provided. The RUD instrument was developed to capture the use of resources by demented patients in a clinical trial setting, which in a further step can be calculated into costs.
Costs of formal care (Utilization of Medical and Nursing services) | 6 months after baseline assessment
  For the health economic evaluation the FIMA (Questionnaire for Health-Related Resource Use in an Elderly Population, Seidl et al. 2015) will be used to determine the supply costs and the formal care provided.
Caregiver Burden (Zarit) | 6 months after baseline assessment
  Caregiver burden will be assessed by using the Zarit Burden Inventory (Zarit, 1980). The instrument consists of 22 items. The result of the instrument is a sum between 22 and 88 - higher results indicate a higher subjective level of burden.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hoffmann, MD, MPH, Prof., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (5):
- Germany (5):
  - MEDIS Ärztenetz medizinischer Versorgung Südbrandenburg, Elsterwerda, Brandenburg
  - GNEF Gesundheitsnetz Frankfurt am Main, Frankfurt am Main, Hesse
  - Demenz-Netzwerk Uckermark e.V., Prenzlau, Mecklenburg- Western Pommerania
  - HaffNet Management GmbH, Ueckermünde, Mecklenburg- Western Pommerania
  - DZNE, Greifswald, Mecklenburg-Vorpommern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichler T, Thyrian JR, Hertel J, Richter S, Wucherer D, Michalowsky B, Teipel S, Kilimann I, Dreier A, Hoffmann W. Unmet Needs of Community-Dwelling Primary Care Patients with Dementia in Germany: Prevalence and Correlates. J Alzheimers Dis. 2016;51(3):847-55. doi: 10.3233/JAD-150935. PMID 26890767
- [Background] van der Roest HG, Meiland FJ, Comijs HC, Derksen E, Jansen AP, van Hout HP, Jonker C, Droes RM. What do community-dwelling people with dementia need? A survey of those who are known to care and welfare services. Int Psychogeriatr. 2009 Oct;21(5):949-65. doi: 10.1017/S1041610209990147. Epub 2009 Jul 15. PMID 19602305
- [Background] Michalowsky B, Eichler T, Thyrian JR, Hertel J, Wucherer D, Laufs S, Flessa S, Hoffmann W. Medication cost of persons with dementia in primary care in Germany. J Alzheimers Dis. 2014;42(3):949-58. doi: 10.3233/JAD-140804. PMID 25125471
- [Background] Reynolds T, Thornicroft G, Abas M, Woods B, Hoe J, Leese M, Orrell M. Camberwell Assessment of Need for the Elderly (CANE). Development, validity and reliability. Br J Psychiatry. 2000 May;176:444-52. doi: 10.1192/bjp.176.5.444. PMID 10912220
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Wimo A, Jonsson L, Zbrozek A. The Resource Utilization in Dementia (RUD) instrument is valid for assessing informal care time in community-living patients with dementia. J Nutr Health Aging. 2010 Oct;14(8):685-90. doi: 10.1007/s12603-010-0316-2. PMID 20922346
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Derived] Radke A, Michalowsky B, Kleinke F, Platen M, Scharf A, Pfaff M, Buchholz M, Muhlichen F, Penndorf P, Schade S, Dombrowski J, Lerch PEM, Reber KC, Austenat-Wied M, Martens C, van den Berg N, Hoffmann W. Efficacy and cost-effectiveness of extended nursing roles in dementia care: Results of the cluster-randomized trial InDePendent. Alzheimers Dement. 2025 Oct;21(10):e70727. doi: 10.1002/alz.70727. PMID 41143334
- [Derived] Scharf A, Michalowsky B, Radke A, Kleinke F, Schade S, Platen M, Buchholz M, Pfaff M, Iskandar A, van den Berg N, Hoffmann W. Identifying and Addressing Unmet Needs in Dementia: The Role of Care Access and Psychosocial Support. Int J Geriatr Psychiatry. 2025 Apr;40(4):e70066. doi: 10.1002/gps.70066. PMID 40148225
- [Derived] Scharf A, Kleinke F, Michalowsky B, Radke A, Pfitzner S, Muhlichen F, Buchholz M, van den Berg N, Hoffmann W. Sociodemographic and Clinical Characteristics of People Living with Dementia and Their Associations with Unmet Healthcare Needs: Insights from the Baseline Assessment of the InDePendent Study. J Alzheimers Dis. 2024;99(2):559-575. doi: 10.3233/JAD-231173. PMID 38669533
- [Derived] Kleinke F, Michalowsky B, Radke A, Platen M, Muhlichen F, Scharf A, Mohr W, Penndorf P, Bahls T, van den Berg N, Hoffmann W. Advanced nursing practice and interprofessional dementia care (InDePendent): study protocol for a multi-center, cluster-randomized, controlled, interventional trial. Trials. 2022 Apr 11;23(1):290. doi: 10.1186/s13063-022-06249-1. PMID 35410437